CLINICAL TRIAL: NCT06696092
Title: A Single Arm, Open Label, Multi-Center Study Evaluating the Efficacy and Safety of WoundClot Surgical
Brief Title: Safety and Efficacy of WoundClot Surgical
Acronym: WCS-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Core Scientific Creations Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSC-CAL-PRO-001
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Surgical Bleeding
Keywords: hemostat; hemostasis; WoundClot; bleeding
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WoundClot Surgical (Experimental): If the pre- and intra-operative eligibility criteria are fulfilled, WoundClot Surgical will be applied to the index bleeding site and success in achieving hemostasis will be evaluated within 5 minutes following the application.
  Interventions: Device: Hemostatic Agent

INTERVENTIONS:
Device: Hemostatic Agent — WoundClot Surgical may be used in a single target bleeding site of each subject.

SUMMARY:
The goal of this clinical trial is to verify that WoundClot Surgical helps stop bleedings which may occur during surgery. It will also help learn more about the safety of WoundClot Surgical. The main questions this clinical trial aims to answer are:

What is the rate at which WoundClot Surgical helps resolve bleeding after it is applied to a site of a bleeding during surgery? How long does it take from the moment WoundClot Surgical is applied to a site of a bleeding during surgery until the bleeding is resolved? What medical problems do participants have if WoundClot Surgical is applied to a site of a bleeding during surgery?

There is a single treatment group in this study and, if a participant is enrolled (ie, gives consent to participate, meets all conditions for study entry, and experiences a bleeding during the surgery), WoundClot Surgical will be applied to the site of bleeding. The enrolled participants will also need to visit the clinic 8 weeks (± 3 days) after the surgery for checkups.

DETAILED DESCRIPTION:
Following provision of consent, the prospective subjects will be screened for eligibility to participate in the study (Visit 1). Screening procedures and evaluations will include laboratory analyses of complete blood count, serum chemistry, coagulation parameters, and a pregnancy test. Medical history and concomitant medications will be recorded. A physical examination will be conducted, and vital signs will be taken.

Once initial eligibility is confirmed, subjects will be scheduled for the procedure for which they are indicated (Visit 2). If the intra-operative eligibility criteria are fulfilled, WoundClot Surgical will be used (study intervention). Time to hemostasis and any additional surgical and non-surgical intervention(s) or reintervention(s), for persistent or recurrent bleeding, respectively, will be recorded.

Two follow-up visits will be conducted, as part of the planned protocol procedures - on the day after the procedure (Visit 3; if the subject is released from the facility on the same day, this Visit will be conducted prior to the release) and 8 weeks ± 3 days after the procedure (Visit 4; last study Visit). Any additional intervention(s) or reintervention(s) for recurrent bleeding and complications of the initial intervention, whether deemed related to the study intervention (device and/or procedure) or not, will be recorded during every study Visit, planned or unscheduled, starting after Visit 2.

Administration of blood products at any time after the study intervention and before end of study will be captured.

Any device deficiencies and any adverse events, whether deemed related to the study device and/or procedure or not, will be recorded at every study Visit, planned or unscheduled.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric, including newborn (from birth to 1 month of age), or adult (aged 80 or below) patient.
2. Undergoing elective (non-emergency), open or laparoscopic soft tissue dissection, vascular, spinal, thyroid, breast, or gastrointestinal surgery, or hepatic resection.

   NOTE: for this study, soft tissue dissection may be part of:

   abdominoplasty, lower anterior resections, abdominal perineal resection, distal pancreatectomy, esophagectomy, skin graft donor site in burn patients, and mastectomy.
3. Indicated for use of topical mechanical hemostat due to mild to moderate bleeding.
4. Has not received transfusion of blood or blood products between screening and study intervention.
5. Has a target bleeding site that is identifiable and has an approximate surface area of less than or equal to 100 cm^2.
6. Has last pre-study-intervention hematology and biochemistry values within the following limits:

   1. hemoglobin ≥ 8 g/dL (g/100 mL)
   2. platelets ≥ 150 x 10^9/L (x 10^3/mm^3)
   3. white blood cells (WBC) ≥ 3.0 x 10^9/L (x 10^3/mm^3)
   4. absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L (x 10^/mm^)
   5. serum creatinine < 1.5 mg/dL
   6. aspartate aminotransferase (AST) < 1.5 x ULN (upper limit of norm)
   7. alanine aminotransferase (ALT) < 1.5 x ULN
   8. alkaline phosphatase (ALP) < 1.5 x ULN
7. Willing and able to return for the required follow-up visits following study enrollment.
8. If able to reproduce, agrees to use a medically accepted form of contraception from the time of consent to completion of all follow-up study visits when engaging in heterosexual intercourse.
9. Signed informed consent.

Exclusion Criteria:

1. If female and of child-bearing potential, has positive pregnancy test during screening and/or is breast-feeding.
2. Participation in another interventional study.
3. Febrile illness within 7 days of study intervention.
4. History of coagulopathy or intra-procedural coagulopathy prior to study intervention.
5. Intra-operative complications requiring resuscitation.
6. Radiofrequency coagulation, other than focal radiofrequency ablation of vessels, of the target bleeding site prior to study intervention.
7. Application of topical hemostat to the target bleeding site prior to study intervention.
8. Known hypersensitivity to carboxymethyl cellulose or compounds containing it or its salts.
9. In patients undergoing vascular surgery where heparin use is required, history of heparin-induced thrombocytopenia.
10. Prisoners.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-10-02 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Rate of clinically-successful hemostasis | Within 5 minutes of application of WoundClot Surgical
  Proportion, in percent, of subjects with clinically-successful hemostasis at the target bleeding site within 5 minutes of applying WoundClot Surgical.

SECONDARY OUTCOMES:
Time to hemostasis | Within 5 minutes of application of WoundClot Surgical
  Time, in seconds, to clinically-successful hemostasis at the target bleeding site, from the treatment application start to the achievement or hemostasis.

CONTACTS AND LOCATIONS:
Locations (8):
- Romania (8):
  - Spitalul Municipal Campina Sectia Clinica Chirurgie, Câmpina, Prahova
  - Spitalul Sf. Constantin Brasov Sectia Chirurgie Generala, Brasov
  - Spitalul Clinic de Urgenta Chirurgie Plastica Reparatorie si Arsuri, Sectia Chirurgie Plastica Microchirugie Reconstructiva II, Bucharest
  - Spitalul Clinic de Urgenta Bucuresti Secția Clinică Chirurgie III, Bucharest
  - Spitalul Clinic de Urgență "Bagdasar Arseni" Bucuresti Secția Chirurgie Generala, Bucharest
  - Spitalul Clinic de Urgență "Bagdasar Arseni" Bucuresti Secția Chirurgie plastica si microchirurgie reconstructiva, Bucharest
  - Spitalul Clinic de Urgență "Bagdasar Arseni" Bucuresti Secția Neurochirurgie II, Bucharest
  - Spitalul Clinic de Urgenta Targu-Mures Clinica de Chirurgie si Ortopedie Pediatrica, Târgu Mureş

IPD SHARING:
Plan to Share IPD: No
Commercial study sponsor